CLINICAL TRIAL: NCT00432354
Title: An Open Labeled Pilot Study of Atorvastatin in Systemic Lupus Erythematosus
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DTCRD 96-03
Record Dates: First submitted 2007-02-06; First posted 2007-02-07 (Estimated); Last update posted 2007-03-20 (Estimated); Status verified 2007-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: statin; systemic lupus erythematosus; microcirculation
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Atorvastatin

INTERVENTIONS:
Drug: atorvastatin

SUMMARY:
The aim of this study is to to determine whether atorvastatin 40mg per day is effective in the treatment of SLE.

DETAILED DESCRIPTION:
Background: Statins are lipid-lower agents with pleiotropic effects. Beyond the traditional effect as inhibitors of 3-hydroxy-3methylglytaryl coenzyme A (HMG-CoA) reductase, it has anti-inflammatory and immunomodulatory properties. The administration of atorvastatin to lupus-prone model NZB/W F1 mice results in a significant reduction in serum IgG anti-dsDNA Abs and decreased proteinuria. In a pilot study with three patients with SLE, simvastatin induced rapid and significant reduction in proteinuria levels. However, further randomized double-blinded placebo-controlled study is pending.

Objective: The goal of this study was to evaluate the clinical efficacy and laboratory effect of atorvastatin in SLE.

Methods: Forty patients with SLE will randomize in two groups to receive atorvastatin or not as an adjuvant to immunosuppressive agent therapy. Patients who received atorvastatin for 6 months will stop atorvastatin for 8 weeks as a washout period. We will cross over the placebo and experimental groups, then given atorvastatin for another 6 months. Primary outcome is improvement of lupus disease status measured by SLEDAI and microcirculation improvement via nailfold capillaroscopy.

ELIGIBILITY:
Inclusion Criteria:

1. 16-80 years of age, fulfilling ACR criteria for the classification of SLE (no limit on disease duration)
2. Active disease status including (1) active nephritis with moderate proteinuria (between 1.0gm/day and 2.5gm/day) despite ongoing immunosuppressive therapy or (2) moderate active extra-renal component of the SLEDAI score in the range of 3 to 10. The SLE-DAI score should have been stable for at least two weeks prior to screening.
3. The type and number immunosuppressive agents were not changed in recent one months

Exclusion Criteria:

1. inability to give informed consent;
2. myositis (CK>3×normal value);
3. dialysis or serum creatinin>2.5mg/dL;
4. abnormal liver function (ALT>3×normal value);
5. pregnant or breastfeeding;
6. life-threatening illness that would interfere with ability to complete the study;
7. current drug or alcohol abuse
8. Already under statin therapy
9. Active SLE disease need added new immunosuppressive agent or increased current drug dosage for more than 50%.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2007-03; Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
The primary outcome was the change in SLE-DAI, a validated composite disease activity score.

SECONDARY OUTCOMES:
The secondary endpoint was the improvement of microcirculation evaluated by Raynaud's condition score and nailfold capillaroscopy in the beginning and end of the atorvastatin.

CONTACTS AND LOCATIONS:
Overall Officials: Ning-Sheng Lai, MD., Ph.D., Study Chair — Vice President of Buddhist Dalin Chi Tzu General Hospital
Locations (2):
- Taiwan (2):
  - Dalin Tzu Chi General Hospital, Chiayi City, Chia-yi
  - Buddhist Dalin Tzu Chi General Hospital, Chiayi City

REFERENCES:
- [Background] Kiss E, Soltesz P, Der H, Kocsis Z, Tarr T, Bhattoa H, Shoenfeld Y, Szegedi G. Reduced flow-mediated vasodilation as a marker for cardiovascular complications in lupus patients. J Autoimmun. 2006 Dec;27(4):211-7. doi: 10.1016/j.jaut.2006.09.008. Epub 2006 Nov 7. PMID 17088047
- [Result] McCarey DW, McInnes IB, Madhok R, Hampson R, Scherbakov O, Ford I, Capell HA, Sattar N. Trial of Atorvastatin in Rheumatoid Arthritis (TARA): double-blind, randomised placebo-controlled trial. Lancet. 2004 Jun 19;363(9426):2015-21. doi: 10.1016/S0140-6736(04)16449-0. PMID 15207950